CLINICAL TRIAL: NCT04636788
Title: Diagnostic and Prognostic Values of EUS-FNA Specimens and Circulating Exosomal Small RNA in Patients With Pancreatic Cancer
Brief Title: Circulating Extracellular Exosomal Small RNA as Potential Biomarker for Human Pancreatic Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Bin Cheng, Professor, Huazhong University of Science and Technology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: E-sR2020
Record Dates: First submitted 2020-11-04; First posted 2020-11-19 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-11

CONDITIONS: Pancreas Adenocarcinoma
Keywords: exosome; snoRNA; endoscopic ultrasound; liquid biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- pancreatic cancer group (Other): pancreatic cancer, anticipated participants: 68
  other pancreatic lesions including MCN, SCN, IPMN, SPN without malignant pathological finding chronic pancreatitis cholangiocarcinoma healthy control anticipated participants: 34
  Interventions: Procedure: Venous sampling

INTERVENTIONS:
Procedure: Venous sampling — venous sampling of 12ml

SUMMARY:
This study is for the verification of biomarkers for pancreatic cancer treatment using small RNA liquid biopsy, combined with EUS-FNA tissues.

DETAILED DESCRIPTION:
CA19-9 is the FDA approved biomarker for the diagnosis of pancreatic cancer. However, the specificity of CA19-9 to differentiate between pancreatic cancer, cholangiocarcinoma, or other pancreatic lesions is not satisfying enough.

Tumor cells secret abundant exosomes in the early stage. Circulating tumor cells are detected mainly in the advanced stage. Meanwhile, the role of non-coding RNA draws more and more attention in tumor area. Exosomes protect inside RNA from plasma RNase. Compared with long RNA, small RNA, including miRNA, snoRNA, tRNA, piRNA could exist more stably.

By means of next-generation sequencing, we look forward to finding new exosomal small RNA biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* age >18
* pancreatic cancer patients
* pancreatic lesions other than PAAD
* chronic pancreatitis
* cholangiocarcinoma

Exclusion Criteria:

* diagnosed with other pathological types of cancer
* treated with chemo/radio/surgery previously

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-11-01 (Estimated); Study Completion 2022-11-01 (Estimated)

PRIMARY OUTCOMES:
senstivity | up to 8 weeks
  sensitivity of exo-sRNA
specificity | up to 8 weeks
  specificity of exo-sRNA to differentiate between PAAD and other benigh or malignant pancreatic occupying lesions

SECONDARY OUTCOMES:
survival time | up to 18 months
  relationship between expression level of chosen exosomal RNA and patients' survival time in PAAD group

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital, Tongji Medical College, HUST, Wuhan, Hubei, China